CLINICAL TRIAL: NCT03008551
Title: The Effect of Empagliflozin Versus Metformin on Hormonal, Metabolic and Cardiovascular Risk Factors in Patients With Polycystic Ovary Syndrome (PCOS) - a Randomised Open-label Parallel Study.
Brief Title: Empagliflozin vs Metformin in PCOS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Version 3.0
Record Dates: First submitted 2016-12-28; First posted 2017-01-02 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — empagliflozin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empagliflozin group (Experimental): Each participant will receive empagliflozin 25mg daily for 3 months
  Interventions: Drug: Empagliflozin
- Metformin group (Active Comparator): Each participant will receive metformin 1500mg daily for 3 months
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Empagliflozin — Each participant will receive empagliflozin 25mg daily for 3 months.
  Other Names: Jardiance
  Arms: Empagliflozin group
Drug: Metformin — Each participant will receive metformin 1500mg daily for 3 months.
  Other Names: Glucophage SR
  Arms: Metformin group

SUMMARY:
This a randomised open-label parallel study involving women with polycystic ovary syndrome (PCOS). The patients will be randomised either to metformin 1500mg or empagliflozin 25mg daily for three months. The aim of the study is to examine the effect of empagliflozin on hormonal, metabolic and cardiovascular risk markers and quality of life in women with PCOS.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is a very common condition in women that may present with irregular periods, excessive hair growth on the face and body, acne and cysts in the ovaries. PCOS is also associated with increased risk of problems later in life like diabetes, high cholesterol levels and heart disease.

In this study, a medication named Empagliflozin will be tested. Empagliflozin belongs to a class of medicines known as SGLT-2 inhibitors. SGLT-2 stands for sodium glucose co-transporter 2. Empagliflozin, in simple terms, helps in reducing high blood glucose levels by increasing the amount of glucose passed in your urine. This medicine is usually used in patients with type 2 diabetes and has led to improved blood pressure and weight loss in addition to improving blood glucose levels.

We want to give Empagliflozin to women with PCOS to see its effect on hormones related to PCOS and the risk factors for diabetes and heart disease. We will be comparing its effects to metformin (another drug for diabetes) which has already been used in PCOS with very good results.

ELIGIBILITY:
Inclusion Criteria:

1. Women, aged 18-45 years (inclusive), with confirmed diagnosis of PCOS based on Rotterdam criteria.
2. Presence of both irregular periods and biochemical hyperandrogenaemia
3. Body mass index ≥25
4. Negative pregnancy test during screening visit and agree to use barrier contraception during the study period.

Exclusion Criteria:

1. Non-classical 21-hydroxylase deficiency, hyperprolactinaemia, Cushing's disease and androgen-secreting tumours will be excluded by appropriate tests.
2. Confirmed diagnosis of diabetes or pre-diabetes.
3. Ongoing, inadequately controlled thyroid disorder (subjects on thyroid hormone replacement therapy must be on stable dose for at least 3 months before screening day)
4. History or presence of malignant neoplasms within the last 5 years (except basal and squamous cell skin cancer and in-situ carcinoma).
5. History or plan of any form of gastrointestinal tract surgery.
6. History of pancreatitis (Acute or Chronic).
7. Any disorder which in the opinion of the investigator might jeopardize subject's safety.
8. Subjects who are on any of the following medications within 3 months of recruitment:

   * Metformin or other insulin-sensitizing medications (e.g., pioglitazone )
   * Hormonal contraceptives (e.g., birth control pills, hormone-releasing implants, etc.)
   * Anti-androgens (e.g., spironolactone, flutamide, finasteride, etc.)
   * Clomiphene citrate or estrogen modulators such as letrozole
   * GnRH modulators such as leuprolide
   * Minoxidil
9. Female who is pregnant, breast feeding or intended to become pregnant or of child bearing potential not using adequate contraceptive methods.
10. eGFR<60
11. Hypersensitivity to lactose
12. Severe hepatic impairment (ALT >3 times ULN)
13. Women with history of recurrent urinary tract infections.
14. Haematocrit above the upper limit of normal range.
15. Have been involved in another medicinal trial (CTIMP) within the past four weeks.
16. Known hypersensitivity to the Investigational Medicinal Products or any of their excipients.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-08-18 (Actual); Primary Completion 2018-04-02 (Actual); Study Completion 2018-04-02 (Actual)

PRIMARY OUTCOMES:
Endothelial function as measured by RHI (reactive hyperaemia index). | Three months treatment with either empagliflozin 25mg or metformin 1500mg daily
  Endothelial function as measured by RHI (reactive hyperaemia index) will be assessed after three months treatment with either empagliflozin 25mg or metformin S/R 1500mg daily

SECONDARY OUTCOMES:
Inflammatory markers (hsCRP) | Three months treatment with either empagliflozin 25mg or metformin 1500mg daily
  Inflammatory markers (hsCRP) will be assessed after three months treatment with either empagliflozin 25mg or metformin S/R 1500mg daily
Insulin resistance as measured by HOMA (fasting glucose & insulin) | Three months treatment with either empagliflozin 25mg or metformin 1500mg daily
  Insulin resistance as measured by HOMA (fasting glucose & insulin) will be assessed after three months treatment with either empagliflozin 25mg or metformin S/R 1500mg daily
Body weight | Three months treatment with either empagliflozin 25mg or metformin 1500mg daily
  Body weight will be assessed after three months treatment with either empagliflozin 25mg or metformin S/R 1500mg daily
Blood pressure | Three months treatment with either empagliflozin 25mg or metformin 1500mg daily
  Blood pressure will be assessed after three months treatment with either empagliflozin 25mg or metformin S/R 1500mg daily
Lipid profile | Three months treatment with either empagliflozin 25mg or metformin 1500mg daily
  Lipid profile will be assessed after three months treatment with either empagliflozin 25mg or metformin S/R 1500mg daily
Hormonal parameters including free androgen index | Three months treatment with either empagliflozin 25mg or metformin 1500mg daily
  Hormonal parameters including free androgen index will be assessed after three months treatment with either empagliflozin 25mg or metformin S/R 1500mg daily
Endothelial function measured by microparticles | Three months treatment with either empagliflozin 25mg or metformin 1500mg daily
  Endothelial function measured by microparticles will be assessed after three months treatment with either empagliflozin 25mg or metformin S/R 1500mg daily
Quality of life Questionnaire | Three months treatment with either empagliflozin 25mg or metformin S/R 1500mg daily
  Quality of life will be assessed after three months treatment with either empagliflozin 25mg or metformin S/R 1500mg daily

CONTACTS AND LOCATIONS:
Overall Officials: Thozhukat Sathyapalan, MBBS FRCP MD, Principal Investigator — University of Hull/Hull and East Yorkshire Hospitals NHS Trust
Locations (1):
- Michael White Centre for Diabetes and Endocrinology, Hull, East Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Javed Z, Papageorgiou M, Deshmukh H, Rigby AS, Qamar U, Abbas J, Khan AY, Kilpatrick ES, Atkin SL, Sathyapalan T. Effects of empagliflozin on metabolic parameters in polycystic ovary syndrome: A randomized controlled study. Clin Endocrinol (Oxf). 2019 Jun;90(6):805-813. doi: 10.1111/cen.13968. Epub 2019 Apr 2. PMID 30866088